CLINICAL TRIAL: NCT03092349
Title: Effect of SonR Based Stimulation-VECtor OPTimisation in Patients With Chronically Implanted Cardiac Resynchronization Devices
Brief Title: SonR Based Stimulation-VECtor OPTimisation in CRT Patients
Acronym: VECTOPT
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left study site
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZNRW-KA-007_KJG
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vector optimisation — Evaluation of hemodynamically best LV Stimulation vector and device programming according to measurements

SUMMARY:
The primary aim of the present study is to investigate whether the optimisation of LVSV in addition to the optimisation of AV-D and VV-D when using the device-based sensor technology mentioned above results in an improved clinical outcome of CRT. Moreover, noninvasive measurements are intended to evaluate hemodynamic differences between the different stimulation configurations using the Finapres® method.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CRT-D implantation according to guidelines at the time of implantation
* Implanted CRT-D system with SonR sensor technology
* Sinus rhythm
* NYHA class II-IV
* Age ≥ 18 years
* Written informed consent to participate in the study

Exclusion Criteria:

* Patients having received a CRT system without SonR sensor technology
* Patients with an insufficient SonR signal
* Confirmed pregnancy
* Age < 18 years
* Life expectancy < 1 year
* Atrial fibrillation / atrial flutter at the time of enrollment
* Unability to give informed consent
* Participation in another clinical study with active therapeutic arm
* Regular follow-up at the study site from enrolment to 12 months follow up not guaranteed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a CRT-D system providing the possibility of SonR-based optimisation of AV-D and VV-D
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
NT-proBNP decrease (-15%) | 12 months
VO2max (+ ≥0.7 ml/min/kg) | 12 months
NYHA class (improvement by ≥ 1 class) | 12 months
QOL (MLHF), score reduction (-15) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Jürgen Gutleben, MD, Principal Investigator — Clinic for Cardiology, Heart and Diabetes Center North Rhine-Westphalia
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No